CLINICAL TRIAL: NCT04613414
Title: Evaluation of an Early Management Strategy for Obstructive Sleep Apnea: A Randomized Trial
Brief Title: Evaluation of an Early Management Strategy for Obstructive Sleep Apnea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Lung Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB20-1667
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Access to Health Care; Time to Treatment; Treatment Adherence; Quality of Care
MeSH Terms: conditions — Sleep Apnea, Obstructive; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Management (Experimental): Scheduled for sleep physician appointment within 1 month of home sleep apnea test/triage
  Interventions: Other: Early Management
- Usual Care (No Intervention): Scheduled for sleep physician appointment approximately 6 months after home sleep apnea test/triage

INTERVENTIONS:
Other: Early Management — Scheduled for sleep physician appointment within 1 month of home sleep apnea test/triage
  Arms: Early Management

SUMMARY:
The primary objective of this study is to evaluate the effect of more timely care for obstructive sleep apnea (OSA) on adherence to positive airway pressure (PAP) therapy at three months after treatment initiation. The secondary objectives are to determine if earlier care improves the treatment effect of PAP on patient reported sleepiness, quality of life and patient satisfaction. We will also evaluate the impact of shorter wait times on patient engagement in therapy by assessing initial acceptance of PAP therapy, patient activation and self-efficacy with respect to OSA treatment.

The study hypothesis is that the early management strategy will be superior to usual care with respect to the primary outcome of PAP adherence at three months.

ELIGIBILITY:
Inclusion Criteria:

* HSAT ODI >= events/hr and ESS 10 - 15 OR
* HSAT ODI 15 - 30 and ESS 15 or lower

Exclusion Criteria:

* Severe nocturnal hypoxemia on HSAT (mean oxygen saturation by pulse oximetry (SpO2) ≤ 85%)
* Severe hypersomnolence (Epworth Sleepiness Scale score ≥ 16)
* Employed in safety-critical occupation
* Recent motor vehicle collision reported on screening questionnaire (within one year)
* Severe hypertension requiring ≥ three antihypertensive medications
* Recent admission to hospital due to unstable cardiopulmonary disease (within 30 days)
* Upcoming major surgery (within six months)
* Prior history of OSA treatment
* Significant co-morbid sleep disorder that would interfere with PAP acclimatization and adherence (e.g., severe insomnia, restless leg syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive airway pressure adherence | 3 months after treatment initiation
  Mean number of hours of positive airway pressure use per night in the four weeks prior to three month follow-up

SECONDARY OUTCOMES:
Positive airway pressure therapy initiation | 1 week after sleep physician visit
  Proportion of patients who initiate positive airway pressure therapy
Adherent to positive airway pressure | 3 months after treatment initiation
  Proportion of patients using positive airway pressure therapy for at least four hours per night on at least 70% of nights during the four weeks prior to the three-month follow-up
Sleepiness | 3 months after treatment initiation
  Change in Epworth Sleepiness Scale score from baseline to three months. Scale is from 0-24 with higher scores indicating greater sleepiness
General health-related quality of life: Change in EuroQoL-5D-3L | 3 months after treatment initiation
  Change in EuroQoL-5D-3L index score (0-1, higher scores indicating greater quality of life), dimensions (problem vs no problem) and visual analogue score (0-100, higher score indicating greater quality of life) from baseline to three months
Disease-specific health-related quality of life: Change in Sleep Apnea Quality of Life Index | 3 months after treatment initiation
  Change in Sleep Apnea Quality of Life Index from baseline to three months. Scale includes four domains scored from 1-7, with higher scores indicating greater quality of life. The overall score is the average from the four domains
Patient satisfaction: Visit-Specific Satisfaction Instrument total score | 3 months after treatment initiation
  Visit-Specific Satisfaction Instrument total score compared between groups at baseline and after three months of PAP therapy. Scale includes 9 questions rated from 1-5. Total score is between 9-45 with higher scores indicating greater satisfaction
Patient activation | 3 months after treatment initiation
  Change in Patient Activation Measure score from baseline to three months. Scale is from 0-100 with higher scores indicating greater activation
Patient activation level | 3 months after treatment initiation
  Change in patient activation level (based on Patient Activation Measure) from baseline to three months. Scale is from 0-100. Participants are classified from activation level 1-4 based on overall score, with higher level indicating greater activation
Self-efficacy: Self-Efficacy Measure for Sleep Apnea score | 3 months after treatment initiation
  Self-Efficacy Measure for Sleep Apnea score compared between groups at baseline and after three months of PAP therapy. There are 3 subscales (risk perception, outcome expectancies, treatment self-efficacy), each scored from 1-4 with higher scores indicating greater self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Pendharkar, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre Sleep Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared upon completion of data sharing agreement
Time Frame: Data will be available 1 year after initial results are published.
Access Criteria: Please contact principal investigator with study proposal